CLINICAL TRIAL: NCT02037646
Title: Evaluating the Effectiveness of Screening Strategies Using Quantitative Versus Qualitative Fecal Immunochemical Test (FIT) to Prioritize Urgency of Colonoscopy Referral - a Randomized Controlled Trial Protocol
Brief Title: Quantitative Versus Qualitative Fecal Immunochemical Tests (FIT) to Prioritize Urgency of Colonoscopy Referral
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 926.24
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Screening; Fecal occult blood; Fecal immunochemical test; Qualitative; Quantitative
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy; Costs and Cost Analysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Qualitative fecal immunochemical test (Other): Stool samples will be tested with the qualitative fecal immunochemical test (qFIT), and will be stratified for colonoscopy as follows:
  >200 ng/dL - colonoscopy with one month 100-200 ng/dL - colonoscopy as per waiting list <100 ng/dL - no colonoscopy
  Cost analysis, anxiety scores and patient satisfaction scores will be calculated for all patients.
  Interventions: Other: Qualitative fecal immunochemical test; Procedure: Colonoscopy; Other: Cost analysis; Other: Anxiety scores; Other: Patient satisfaction scores
- Quantitative fecal immunochemical test (Other): Stool samples will be tested with the quantitative fecal immunochemical test (FIT), and will be scheduled for colonoscopy as follows:
  Positive - colonoscopy as per waiting list Negative - no colonoscopy
  Cost analysis, anxiety scores and patient satisfaction scores will be calculated for all patients.
  Interventions: Other: Quantitative fecal immunochemical test; Procedure: Colonoscopy; Other: Cost analysis; Other: Anxiety scores; Other: Patient satisfaction scores

INTERVENTIONS:
Other: Qualitative fecal immunochemical test — This test measures the amount of blood within the submitted stool specimen
  Arms: Qualitative fecal immunochemical test
Other: Quantitative fecal immunochemical test — This test detects presence or absence of blood within a submitted stool specimen.
  Arms: Quantitative fecal immunochemical test
Procedure: Colonoscopy — Patients with positive tests will be subjected to colonoscopy to determine presence or absence of advanced colorectal neoplasms.
Other: Cost analysis — Data on direct and indirect costs to patient and institution will be collected at each patient visit related to screening.
Other: Anxiety scores — Hospital Anxiety and Depression Scale (HADS) questionnaire
Other: Patient satisfaction scores — A 5-point patient satisfaction score will be documented at each patient visit related to screening.

SUMMARY:
The main aim of this study is to determine whether there is a difference in time to diagnosis of advanced colorectal neoplasms using quantitative Fecal Immunochemical Tests (FIT) to prioritize referral for colonoscopy (intervention) compared to usual care (qualitative FIT and appointment-based referral).

DETAILED DESCRIPTION:
It is hypothesized that quantitative FIT will enable faster detection of advanced neoplasms compared to qualitative FIT.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 years and above

Exclusion Criteria:

* Lower gastrointestinal tract symptoms such as diarrhoea, constipation, per rectal bleeding
* Personal history of colorectal tumour or cancer
* Family history of familial adenomatous polyposis or hereditary non-polyposis colorectal cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to diagnosis of advanced colorectal neoplasms | 40-90 days from the time of enrolment
  Measured as number of days from the time of enrolment until histological diagnosis of a colorectal neoplasm

SECONDARY OUTCOMES:
Analysis of screening costs | Up to 90 days following enrolment
  Total costs incurred as a result of the screening process
Patient anxiety levels | Up to 90 days after enrolment
  As measured by the Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: April C Roslani, MBBCh, Principal Investigator — University of Malaya Medical Centre
Locations (1):
- University of Malaya Medical Centre, Kuala Lumpur, Malaysia